CLINICAL TRIAL: NCT06276114
Title: Comparison of Intravascular Coronary Lithotripsy and Excimer Laser Coronary Atherectomy for Severe Stent Underexpansion: the Multicenter IVL- ELCA DRAGON Registry
Brief Title: IVL vs ELCA for Stent Underexpantsion (IVL-ELCA DRAGON)
Acronym: DRAGON
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Prof. Ass., Medical University of Silesia
Other Study IDs: 07
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Calcification; Intravascular Lithotripsy; Excimer Laser-coronary Atherectomy; Stent Restenosis; Stent Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consecutive patients with stent underexpantsion treated with IVL
  Interventions: Device: Stent Underexpansion
- Consecutive patients with stent underexpantsion treated ELCA
  Interventions: Device: Stent Underexpansion

INTERVENTIONS:
Device: Stent Underexpansion — Stent underexpansion was diagnosed as stent expansion of <80% assessed with intravascular imaging.

SUMMARY:
The IVL- ELCA DRAGON Registry is a multicenter study that enrolled consecutive patients with stent underexpansion treated with IVL ora ELCA in high-volume PCI centers.

The primary efficacy endpoint was device success (technical success with a final stent expansion ≥ 80%). Thirty days device-oriented composite endpoint (DOCE: cardiac death, target lesion revascularization, or target vessel myocardial infarction) was the secondary endpoint.

ELIGIBILITY:
Stent underexpansion as stent expansion of <80% assessed with intravascular imaging (minimum in-stent lumen area divided by average reference lumen area x100%).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with underexpanded coronary stent were included regardless of time since stent implantation. Patients who did not undergo intravasuclar imaging during PCI were excluded.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was device success | During procedure
  Technical success with a final stent expansion ≥80%.

SECONDARY OUTCOMES:
Device-oriented composite endpoint (DOCE) | Thirty days
  cardiac death, target lesion revascularization, or target vessel myocardial infarction

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (2):
  - Unit of Structural Interventional Cardiology, Department of Clinical and Experimental Medicine, Careggi University Hospital, Florence
  - Fabrizio D'Ascenzo, Turin
- Poland (18):
  - Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok
  - First Department of Cardiology, Medical University of Gdansk, Gdansk, Poland, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Jacek Legutko, Krakow
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow
  - 1st Military Hospital in Lublin, Lublin, Poland, Lubin
  - Department of Cardiology, Copper Health Centre (MCZ), Lubin
  - Clinical Department of Interventional Cardiology, Medical University of Lublin, Lublin
  - Department of Cardiology, University Hospital, Institute of Medical Sciences, Opole
  - Department of Cardiology, Poznan University of Medical Sciences, Poznan
  - Department of Cardiology, The Ministry of Internal Affairs and Administration Hospital, Rzeszow, Rzeszów
  - 1st Department of Cardiology, Medical University of Warsaw, Warsaw
  - Department of Cardiology and Internal Diseases, Military Institute of Medicine, Warsaw
  - Department of Interventional Cardiology and Angiology, National Institute of Cardiology, Warsaw, Poland, Warsaw
  - Department of Invasive Cardiology, Centre of Postgraduate Medical Education, Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Department of Invasive Cardiology, Wejherowo, Wejherowo
  - Centre for Heart Disease, University Hospital Wroclaw Department of Heart Disease, Wroclaw Medical University, Wroclaw
  - Third Department of Cardiology, Medical University of Katowice, Zabrze

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wanha W, Tomaniak M, Wanczura P, Bil J, Januszek R, Wolny R, Opolski MP, Kuzma L, Janas A, Figatowski T, Gasior P, Milewski M, Roleder-Dylewska M, Lewicki L, Kulczycki J, Wlodarczak A, Tomasiewicz B, Iwanczyk S, Sacha J, Koltowski L, Dziarmaga M, Jaguszewski M, Kralisz P, Olajossy B, Sobieszek G, Dyrbus K, Lebek M, Smolka G, Reczuch K, Gil RJ, Dobrzycki S, Kwiatkowski P, Rogala M, Gasior M, Ochala A, Kochman J, Witkowski A, Lesiak M, D'Ascenzo F, Bartus S, Wojakowski W. Intravascular Lithotripsy for the Treatment of Stent Underexpansion: The Multicenter IVL-DRAGON Registry. J Clin Med. 2022 Mar 23;11(7):1779. doi: 10.3390/jcm11071779. PMID 35407387